CLINICAL TRIAL: NCT06127043
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Rosnilimab in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: A Study of Efficacy and Safety of Rosnilimab in Subjects With Moderate to Severe Ulcerative Colitis (ROSETTA)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AnaptysBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANB030-204 ROSETTA
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis
Keywords: Rosnilimab; ANB030; PD-1 agonist; ROSETTA
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rosnilimab SC Dose 1 (Experimental): This arm will receive High dose Rosnilimab SC
  Interventions: Drug: Rosnilimab
- Rosnilimab SC Dose 2 (Experimental): This arm will receive low dose Rosnilimab SC
  Interventions: Drug: Rosnilimab
- Placebo (Placebo Comparator): This arm will receive Placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosnilimab — PD-1 agonist antibody
  Other Names: ANB030
  Arms: Rosnilimab SC Dose 1; Rosnilimab SC Dose 2
Drug: Placebo — Administered via SC
  Arms: Placebo

SUMMARY:
ROSETTA STUDY: This study will evaluate the safety, tolerability, and efficacy of Rosnilimab in subjects with moderate to severe ulcerative colitis (UC)

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy, safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of rosnilimab in subjects with moderate to severe ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18
* Participants with a clinical diagnosis of UC for prior to Day 1
* Subject has moderate to severe, active UC, defined as a mMS ≥ 5 with an endoscopy subscore ≥2
* Subject has had a surveillance colonoscopy that did not detect potential dysplasia or colon cancer performed within 1 year of Day 1.
* Subject has a history of an inadequate response, loss of response, or intolerance to any combination of at least 2 UC therapy classes defined as, but not limited to, aminosalicylates, corticosteroids, immunomodulators, calcineurin inhibitors, or advanced UC therapies (e.g., biologics, JAK inhibitors, oral S1P receptor modulators, etc.)

Exclusion Criteria:

* Subject has a diagnosis of Crohn's disease or indeterminate colitis.
* Subject has a diagnosis of fulminant colitis and/or toxic megacolon.
* Subject has a history of an inadequate response, loss of response, or intolerance to any combination of 3 or more advanced UC therapy classes but not limited to, 1) anti-TNF antibodies (e.g., adalimumab, golimumab, infliximab), 2) other biologics (e.g., ustekinumab, vedolizumab), 3) oral JAK inhibitors (e.g., tofacitinib, upadacitinib), and 4) oral S1P receptor modulators (e.g., ozanimod).
* Subject has disease limited to the rectum (ulcerative proctitis)
* Subject has a history of colectomy (total or subtotal), ileoanal pouch, Kock pouch, or ileostomy or is planning bowel surgery.
* The subject had prior exposure to a PD-1 or PD-L1 agonist, antagonist, or modulator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean change in modified Mayo Score (mMs) from Baseline to Week 12 | Baseline to Week 12
  The mMS is an endoscopic and clinical scale, which ranges in scores from 0-9, with higher numbers indicating increased disease severity. It is used to assess UC disease activity. It consists of three subscores: RBS, SFS and an endoscopy subscore.

SECONDARY OUTCOMES:
Proportion of subjects achieving clinical remission at Week 12 | Baseline to Week 12
  Defined as a mMS ≤ 2, with a stool frequency subscore (SFS) ≤ 1, RBS=0, and endoscopic subscore ≤ 1 without friability.
Proportion of subjects showing endoscopic treatment improvement at Week 12 | Baseline to Week 12
  Defined as an endoscopy subscore ≤ 1 without friability.
Proportion of subjects achieving a clinical response at Week 12 | Baseline to Week 12
  Defined as a decrease from Baseline in mMS ≥ 2 points and ≥ 30% with a decrease from Baseline in RBS ≥ 1 point or an absolute RBS ≤ 1.

CONTACTS AND LOCATIONS:
Overall Officials: Zurab Machaidze, MD, Study Director — AnaptysBio, Inc.
Locations (100):
- United States (25):
  - AnaptysBio Investigational Site 10-115, Phoenix, Arizona
  - AnaptysBio Investigational Site 10-117, Garden Grove, California
  - AnaptysBio Investigational Site 10-112, Lancaster, California
  - AnaptysBio Investigational Site 10-129, Lancaster, California
  - AnaptysBio Investigational Site 10-108, San Jose, California
  - AnaptysBio Investigational Site 10-127, Brooksville, Florida
  - AnaptysBio Investigational Site 10-106, Miami, Florida
  - AnaptysBio Investigational Site 10-109, Miami Gardens, Florida
  - AnaptysBio Investigational Site 10-131, Orlando, Florida
  - AnaptysBio Investigational Site 10-123, Orlando, Florida
  - AnaptysBio Investigational Site 10-125, Tampa, Florida
  - AnaptysBio Investigational Site 10-122, Atlanta, Georgia
  - AnaptysBio Investigational Site 10-124, Oak Lawn, Illinois
  - AnaptysBio Investigational Site 10-118, Las Vegas, Nevada
  - AnaptysBio Investigational Site 10-133, Utica, New York
  - AnaptysBio Investigational Site 10-136, Cincinnati, Ohio
  - AnaptysBio Investigational Site 10-120, Norman, Oklahoma
  - AnaptysBio Investigational Site 10-103, Kingsport, Tennessee
  - AnaptysBio Investigational Site 10-104, Dallas, Texas
  - AnaptysBio Investigational Site 10-113, Garland, Texas
  - AnaptysBio Investigational Site 10-135, Georgetown, Texas
  - AnaptysBio Investigational Site 10-134, Lubbock, Texas
  - AnaptysBio Investigational Site 10-130, Southlake, Texas
  - AnaptysBio Investigational Site 10-132, Tyler, Texas
  - AnaptysBio Investigational Site 10-107, Seattle, Washington
- Austria (4):
  - AnaptysBio Investigational Site 12-101, Innsbruck
  - AnaptysBio Investigational Site 12-104, Salzburg
  - AnaptysBio Investigational Site 12-103, Sankt Pölten
  - AnaptysBio Investigational Site 12-102, Vienna
- AnaptysBio Investigational Site 61-102, Sofia, Bulgaria
- Canada (3):
  - AnaptysBio Investigational Site 11-102, London, Ontario
  - AnaptysBio Investigational Site 11-103, Montreal, Quebec
  - AnaptysBio Investigational Site 11-105, Calgary
- Croatia (2):
  - AnaptysBio Investigational Site 74-104, Rijeka
  - AnaptysBio Investigational Site 74-101, Zagreb
- France (3):
  - AnaptysBio Investigational Site 16-102, Nantes
  - AnaptysBio Investigational Site 16-103, Nantes
  - AnaptysBio Investigational Site 16-101, Tours
- Georgia (6):
  - AnaptysBio Investigational Site 59-101, Tbilisi, Georgia
  - AnaptysBio Investigational Site 59-106, Tbilisi
  - AnaptysBio Investigational Site 59-103, Tbilisi
  - AnaptysBio Investigational Site 59-102, Tbilisi
  - AnaptysBio Investigational Site 59-104, Tbilisi
  - AnaptysBio Investigational Site 59-105, Tbilisi
- Germany (8):
  - AnaptysBio Investigational Site 17-107, Berlin
  - AnaptysBio Investigational Site 17-106, Brandenburg
  - AnaptysBio Investigational Site 17-105, Dachau
  - AnaptysBio Investigational Site 17-101, Duisburg
  - AnaptysBio Investigational Site 17-110, Erlangen
  - AnaptysBio Investigational Site 17-108, Hamburg
  - AnaptysBio Investigational Site 17-103, Kiel
  - AnaptysBio Investigational Site 17-109, Ulm
- Italy (11):
  - AnaptysBio Investigational Site 20-112, Bologna
  - AnaptysBio Investigational Site 20-111, Cagliari
  - AnaptysBio Investigational Site 20-110, Catania
  - AnaptysBio Investigational Site 20-108, Legnano
  - AnaptysBio Investigational Site 20-105, Milan
  - AnaptysBio Investigational Site 20-107, Pavia
  - AnaptysBio Investigational Site 20-102, Rozzano
  - AnaptysBio Investigational Site 20-109, San Donato
  - AnaptysBio Investigational Site 20-104, San Giovanni
  - AnaptysBio Investigational Site 20-113, Turin
  - AnaptysBio Investigational Site 20-106, Udine
- AnaptysBio Investigational Site 21-101, Amsterdam, Netherlands
- Poland (19):
  - AnaptysBio Investigational Site 30-108, Bydgoszcz
  - AnaptysBio Investigational Site 30-106, Częstochowa
  - AnaptysBio Investigational Site 30-112, Elblag
  - AnaptysBio Investigational Site 30-102, Katowice
  - AnaptysBio Investigational Site 30-115, Katowice
  - AnaptysBio Investigational Site 30-111, Krakow
  - AnaptysBio Investigational Site 30-123, Krakow
  - AnaptysBio Investigational Site 30-103, Lodz
  - AnaptysBio Investigational Site 30-119, Lodz
  - AnaptysBio Investigational Site 30-114, Lublin
  - AnaptysBio Investigational Site 30-104, Poznan
  - AnaptysBio Investigational Site 30-117, Poznan
  - AnaptysBio Investigational Site 30-120, Poznan
  - AnaptysBio Investigational Site 30-116, Rzeszów
  - AnaptysBio Investigational Site 30-113, Sopot
  - AnaptysBio Investigational Site 30-110, Torun
  - AnaptysBio Investigational Site 30-101, Warsaw
  - AnaptysBio Investigational Site 30-107, Warsaw
  - AnaptysBio Investigational Site 30-109, Warsaw
- Romania (3):
  - AnaptysBio Investigational Site 30-101, Bucharest
  - AnaptysBio Investigational Site 31-103, Cluj-Napoca
  - AnaptysBio Investigational Site 31-102, Timișoara
- Serbia (5):
  - AnaptysBio Investigational Site 58-101, Belgrade
  - AnaptysBio Investigational Site 58-103, Belgrade
  - AnaptysBio Investigational Site 58-104, Belgrade
  - AnaptysBio Investigational Site 58-105, Belgrade
  - AnaptysBio Investigational Site 58-102, Zrenjanin
- Spain (2):
  - AnaptysBio Investigational Site 24-102, Alicante
  - AnaptysBio Investigational Site 24-103, Lleida
- United Kingdom (7):
  - AnaptysBio Investigational Site 27-103, Belfast
  - AnaptysBio Investigational Site 27-102, Cambridge
  - AnaptysBio Investigational Site 27-106, Liverpool
  - AnaptysBio Investigational Site 27-101, London
  - AnaptysBio Investigational Site 27-105, Runcorn
  - AnaptysBio Investigational Site 27-107, Shrewsbury
  - AnaptysBio Investigational Site 27-104, York

IPD SHARING:
Plan to Share IPD: No